CLINICAL TRIAL: NCT07158450
Title: Evaluation of Wearable Sensor-Based Estimation of Left Ventricular Ejection Fraction (LVEF) - Pilot Study
Brief Title: Novel On-body Evaluation of Cardiac Health for Oncology
Acronym: NOECHO
Status: Enrolling by invitation | Type: Observational
Sponsor: Skribe Medical (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: SKR-LVEF-001
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cardiotoxicity; Heart Failure
MeSH Terms: conditions — Cardiotoxicity; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy: No known or suspected cardiac disease
- Borderline LVEF: Known conditions that may predispose to LV dysfunction, but no prior diagnosis of reduced left ventricular ejection fraction
- Reduced LVEF: Known diagnosis of reduced left ventricular ejection fraction

SUMMARY:
The goal of this study is to develop a wearable sensor system that can estimate left ventricular ejection fraction (LVEF), which is a measurement of the heart's function.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an echocardiogram irrespective of participation in this study
* Willing and able to provide informed consent prior to any study-related activity

Exclusion Criteria:

* Have a documented allergy to potential tissue contacting system materials
* Have been diagnosed with one or more of the following cardiac diseases/conditions that distort cardiac activity:

  1. Severe valve disease
  2. Severe right ventricular dilation or dysfunction
  3. Significant arrhythmias or conduction abnormalities
  4. Active ischemia or myocardial infarction within the last 3 months
* Have an active implantable cardiac device
* Have any condition that would cause inaccurate TTE measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) recruited from participating cardiology clinics. Participants are assigned to one of three cohorts by transthoracic echocardiography (TTE): Healthy (no known structural heart disease; LVEF ≥ 55%), Borderline/Possibly reduced LVEF (LVEF 40-54% or clinical concern for decline), and Reduced LVEF (LVEF < 40%). The population is intended to span the full spectrum of systolic function for model training and evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between wearable-derived and transthoracic echocardiography-derived left ventricular ejection fraction estimates | From baseline through study completion (up to 6 months) at each paired assessment
  The primary analysis will compute the correlation coefficient (r) between wearable-derived model estimates of LVEF and transthoracic echocardiography-derived LVEF in the Hold-Out Test Set. The prespecified performance target is r > 0.70.

SECONDARY OUTCOMES:
Clinical accuracy of wearable-derived LVEF compared with echocardiography | From baseline through study completion (up to 6 months) at each paired assessment
  Proportion of predictions within ±5 percentage points of TTE-derived LVEF in the Hold-Out Test Set. Error metrics will be calculated as Mean Absolute Error (MAE) between wearable-derived and TTE-derived LVEF. Differences across subgroups will be tested with ANOVA or Kruskal-Wallis as appropriate. Prespecified performance target: MAE ≤ 5 percentage points.

CONTACTS AND LOCATIONS:
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to proprietary device algorithms and consent restrictions.